CLINICAL TRIAL: NCT04240886
Title: A Phase 2, Open-Label Study to Evaluate the Safety and Efficacy of APX001 in the Treatment of Patients With Invasive Mold Infections Caused by Aspergillus Species or Rare Molds
Brief Title: Open-label Study of APX001 for Treatment of Patients With Invasive Mold Infections Caused by Aspergillus or Rare Molds
Acronym: AEGIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor made a strategic decision to terminate the study, in order to prioritize a randomized comparative Phase 3 trial in the same indication. This decision was not based on any safety concerns
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APX001-202; C4791010 (Other: Alias Study Number); 2019-001386-33 (EudraCT Number)
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Invasive Fungal Infections
Keywords: APX001; APX001A; fosmanogepix; manogepix; aspergillus; aspergillosis; covid; covid19; mold; mould; pulmonary aspergillosis; pulmonary aspergillus; galactomannan; Karius; SARS-CoV-2; fusarium; mucorales; mucor; rhizopus; scedosporium; fungal disease; invasive fungal disease; EORTC
MeSH Terms: conditions — Invasive Fungal Infections; Aspergillosis; COVID-19; Pulmonary Aspergillosis; Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: fosmanogepix (APX001) (Experimental)
  Interventions: Drug: fosmanogepix
- Cohort B: fosmanogepix (APX001) (Experimental)
  Interventions: Drug: fosmanogepix

INTERVENTIONS:
Drug: fosmanogepix — IV and oral fosmanogepix
  Other Names: APX001; E210

SUMMARY:
This is a Phase 2, multicenter study to evaluate APX001 for the treatment of invasive fungal infections caused by Aspergillus spp. or rare molds (eg, Scedosporium spp., Fusarium spp., and Mucorales fungi).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 years or older.
* Patients with proven or probable IMI caused by Aspergillus spp. Patients who present with IMI due to other filamentous fungi (eg, Scedosporium spp., Fusarium spp., and Mucorales fungi such as Mucor spp. or Rhizopus spp.) may also be enrolled.
* Have limited or no treatment options due to documented or anticipated resistance, contraindication, intolerance, or lack of clinical response to SOC antifungal therapy, as advocated by the relevant regional/country treatment guidelines.
* Patients where the Investigator considers that there is a potential advantage of using APX001 over current SOC (eg, broad spectrum of activity, emergence of IMI during antifungal prophylaxis, activity against resistant mold pathogens, IV and PO formulations, favorable DDI profile, favorable hepatic and renal safety profile, wide tissue distribution including brain), and/or where the SOC antifungal therapy carries significant risk of toxicity or treatment failure (eg, DDI risk, safety/toxicity risk, site of infection not accessible by SOC).

Exclusion Criteria:

* Refractory hematologic malignancy.
* Chronic aspergillosis, aspergilloma, or allergic bronchopulmonary aspergillosis.
* Treatment with systemic (PO, IV, or inhaled) mold active antifungal therapy for 120 hours immediately before initial dosing. Note: patients with invasive fungal infection caused by a mold with documented resistance to or lack of coverage by the prior SOC in question, may have received >120 hours prior treatment and remain eligible for the study.
* Evidence of significant hepatic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (15):
- United States (6):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - IP Address : City of Hope Investigational Drug Services (IDS), Duarte, California
  - Duke Department of Pharmacy/Investigational Drug Service (IDS), Durham, North Carolina
  - Duke Medicine Pavilion, Durham, North Carolina
  - Duke University Medical Center (Duke South Clinic), Durham, North Carolina
  - Duke University Medical Center(Duke Hospital), Durham, North Carolina
- Belgium (3):
  - Cliniques Universitaires de Bruxelles Hôpital Erasme - Department of Infectious Diseases, Brussels
  - UZ Leuven - Department of Haematology, Leuven
  - CHU UCL Namur - Mont- Godinne University Hospital - Intensive Care Unit, Yvoir
- Germany (2):
  - Klinikum Neuperlach, Klinik fur Hamatologie und Onkologie, München, Bavaria
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz III, Mainz
- Israel (4):
  - Pharmacy, Haifa
  - Rambam Medical Center, Haifa
  - Pharmacy, Ramat Gan
  - Sheba Medical Center, Tel Hashomer, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodges MR, Tawadrous M, Cornely OA, Thompson GR, Slavin MA, Maertens JA, Dadwal SS, Rahav G, Hazel S, Almas M, Jakate A, Pypstra R. Fosmanogepix for the Treatment of Invasive Mold Diseases Caused by Aspergillus Species and Rare Molds: A Phase 2, Open-Label Study (AEGIS). Clin Infect Dis. 2025 Dec 24;81(5):e302-e309. doi: 10.1093/cid/ciaf185. PMID 40203286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was planned to be conducted in two parallel cohorts: Cohort A included participants with invasive mold infections (IMA) and an exploratory Cohort B was planned to include participants with invasive aspergillus, who had COVID-19 or Influenza A/B. The study was terminated early and no participants were enrolled in Cohort B; hence data is not reported for Cohort B in any section.
Groups:
- APX001 (Fosmanogepix): Cohort A: Eligible participants aged 18 years or older with invasive mold infections (IMI) and limited antifungal treatment options were included in this arm. On Day 1, participants received APX001 1000 milligram (mg) as a loading dose over 3 hours by intravenous (IV) infusion twice daily (BID). On Days 2 and 3, participants received APX001 600 mg as maintenance dose over 3 hours by IV infusion once daily (QD). From Day 4 till end of study treatment, for maintenance dose participants received either APX001 600 mg IV infusion QD over 3 hours or switched to APX001 800 mg orally QD on investigator discretion. Total treatment duration was maximum of 42 days. Participants had a follow-up visit at 4 weeks after last dose of study treatment and a follow-up telephone call was required on Day 84.
Period: Treatment Phase
Arm/Group | APX001 (Fosmanogepix): Cohort A
Started | 21
Completed | 11
Not Completed | 10
Not completed — Death | 4
Not completed — Discontinuation by Subject | 1
Not completed — Adverse Event | 5
Period: Follow-up Phase
Arm/Group | APX001 (Fosmanogepix): Cohort A
Started | 17 (Eligible participants entered follow-up period following discontinuation of study treatment)
Completed | 13
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Discontinuation by Subject | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.38 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died After the First Dose of Study Drug Through Day 42
Description: Percentage of participants who died after first dose in the study through Day 42 were reported in this outcome measure. This outcome measure included all deaths from Day 1 through Day 42.
Time Frame: After first dose on Day 1 through Day 42
Population: The modified Intent-to-Treat (mITT) population included all participants who entered in the study, received at least 1 dose of study drug, and had a diagnosis of proven or probable IMI confirmed by the DRC.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 20
Percentage of participants | 25.0 [12.7 to 41.5]

2. Secondary Outcome: Percentage of Participants With Global Response Based on Data Review Committee (DRC) Assessment at End of Study Drug Treatment (EOST)
Description: Global response was classified as treatment success (complete or partial response [CR or PR]) or treatment failure (stable response [SR], progression of fungal disease [PD], or death) as determined by DRC. CR: survival within prespecified period of observation (PPOB), resolution of all attributable (att) symptoms and signs of disease and radiological (rad) abnormalities, and mycological (myco) evidence of eradication of disease. PR: survival within POB, improvement in att symptoms and signs of disease and rad abnormalities, and evidence of clearance of cultures or reduction of fungal burden. SR: survival within PPOB, minor or no improvement in fungal disease but no evidence of progression based on composite of clinical, rad and myco criteria, PD or death. PD: evidence of progressive fungal disease based on composite of clinical, rad and myco criteria. Death: death during PPOB, regardless of attribution. Data is presented for EOST which could have preceded Day 42 for some participants.
Time Frame: Any day from Day 1 until end of study treatment (any day up to Day 42)
Population: mITT population included all participants who entered in the study, received at least 1 dose of study drug, and had a diagnosis of proven or probable IMI confirmed by the DRC.
Measure: Number; unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 20
Percentage of participants
  CR | 20.0
  PR | 20.0
  SR | 10.0
  PD | 30.0
  Death | 20.0

3. Secondary Outcome: Percentage of Participants With Treatment Success or Treatment Failure for Global Response Based on Data Review Committee (DRC) Assessment at End of Study Drug Treatment (EOST)
Description: Global response was classified as treatment success (CR or PR) or treatment failure (SR, PD or death) as determined by DRC. CR: survival within prespecified POB, resolution of all attributable symptoms and signs of disease and rad abnormalities and myco evidence of eradication of disease. PR: survival within prespecified POB, improvement in attributable symptoms and signs of disease and rad abnormalities and evidence of clearance of cultures or reduction of fungal burden. SR: survival within prespecified POB, minor or no improvement in fungal disease, but no evidence of progression, based on composite of clinical, rad, and myco criteria, PD or death. PD: evidence of PD based on a composite of clinical, rad, and myco criteria. Death: death during prespecified period of evaluation, regardless of attribution. Percentage of participants with treatment success (CR, PR) and treatment failure (SR, PD, death) along with two-sided exact binomial 80% confidence interval is presented.
Time Frame: Any day from Day 1 until end of study treatment (any day up to Day 42)
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 20
Percentage of participants
  Treatment Success | 40.0 [24.9 to 56.7]
  Treatment Failure | 60.0 [43.3 to 75.1]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between first dose of study drug and up to 4 weeks post last dose of study treatment that were absent before treatment or that worsened relative to pretreatment state. An SAE was any untoward medical occurrence that occurred, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; was a congenital anomaly/birth defect and other important medical events. AEs included SAEs and all non-SAEs.
Time Frame: Day 1 up to maximum of 31 days of follow up post last dose of study treatment, where maximum treatment duration was 42 days (maximum up to 73 days)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
Participants
  TEAEs | 21
  SAEs | 13

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Vital Signs
Description: Vital signs included body temperature, blood pressure, heart rate, respiratory rate, and oxygen saturation. Number of participants with clinically significant abnormality in vital signs as judged by investigator were reported in this outcome measure.
Time Frame: as for outcome 4
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
Participants | 5

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Laboratory Test Evaluations
Description: Clinical laboratory assessments included serum chemistry (bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, creatinine, creatine kinase), hematology (including hemoglobin, hematocrit, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils and monocytes), coagulation (including Prothrombin time [PT]/ International normalized ratio [INR]), and urinalysis. Number of participants with clinically significant abnormality in any laboratory parameter as judged by investigator and reported as adverse events were presented.
Time Frame: as for outcome 4
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
Participants | 12

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval, QRS interval, QT interval, QT interval corrected using the Fridericia's formula (QTcF), QT interval corrected using the Bazett's formula (QTcB), RR interval and heart rate. Number of participants with clinically significant abnormal ECG findings as judged by investigator were presented.
Time Frame: as for outcome 4
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
Participants | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical and Neurological Examinations
Description: Physical examination included an assessment of general appearance, skin, eyes, heart, chest, abdomen, and a neurological examination. Components of the neurological examination included cranial nerve, sensory, and motor examination; reflex and gait testing; and coordination assessment. Clinically significant changes were judged by investigator.
Time Frame: as for outcome 4
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
Participants | 3

9. Secondary Outcome: Plasma Concentrations of Fosmanogepix
Time Frame: Days 1, 2, 3, 4, 7: Pre-dose and 3 hours post-dose; Days 6, 13, 14: 3 hours post-dose, Day 15: pre-dose
Population: The Pharmacokinetic (PK) Population included all participants who received any amount of study drug and had evaluable PK data. Here, "Number Analyzed" signifies participants evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | APX001 (Fosmanogepix): Cohort A
Number analyzed (Participants) | 21
nanogram per milliliter
  Day 1: Pre-dose | 0.0 (0.0)
  Day 1: 3 hrs post-dose: number analyzed (Participants) | 18
  Day 1: 3 hrs post-dose | 387.4 (289.6)
  Day 2: Pre-dose: number analyzed (Participants) | 7
  Day 2: Pre-dose | 20.4 (138.1)
  Day 2: 3 hrs post-dose: number analyzed (Participants) | 20
  Day 2: 3 hrs post-dose | 406.4 (202.9)
  Day 3: Pre-dose: number analyzed (Participants) | 6
  Day 3: Pre-dose | 8.6 (184.1)
  Day 3: 3 hrs post-dose: number analyzed (Participants) | 19
  Day 3: 3 hrs post-dose | 486.7 (154.6)
  Day 4: Pre-dose: number analyzed (Participants) | 2
  Day 4: Pre-dose | 2.9 (141.3)
  Day 4: 3 hrs post-dose: number analyzed (Participants) | 2
  Day 4: 3 hrs post-dose | 85.2 (14743.4)
  Day 6: 3 hrs post-dose: number analyzed (Participants) | 2
  Day 6: 3 hrs post-dose | 6.8 (1541.9)
  Day 7: Pre-dose: number analyzed (Participants) | 2
  Day 7: Pre-dose | 9.8 (716.5)
  Day 7: 3 hrs post-dose: number analyzed (Participants) | 7
  Day 7: 3 hrs post-dose | 37.9 (382.3)
  Day 13: 3 hrs post-dose: number analyzed (Participants) | 1
  Day 13: 3 hrs post-dose | 96.4 (NA) — Geometric coefficient of variation could not be calculated as a single participant was analyzed
  Day 14: 3 hrs post-dose: number analyzed (Participants) | 4
  Day 14: 3 hrs post-dose | 706.8 (181.0)
  Day 15: Pre-dose: number analyzed (Participants) | 1
  Day 15: Pre-dose | 0.5 (NA) — Geometric coefficient of variation could not be calculated as a single participant was analyzed

ADVERSE EVENTS:
Time Frame: For adverse events (SAEs and non-SAEs): Day 1 up to maximum of 31 days of follow up post last dose of study treatment, where maximum treatment duration was 42 days (maximum up to 73 days); for all-cause mortality: Throughout the study (Day 1 to Day 84)
Description: Same event may appear as SAE and non-SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | APX001 (Fosmanogepix): Cohort A
All-Cause Mortality (participants affected / at risk) | 9/21
Serious Adverse Events (participants affected / at risk) | 13/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APX001 (Fosmanogepix): Cohort A (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 1
Catheter site infection (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Stenotrophomonas bacteraemia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APX001 (Fosmanogepix): Cohort A (N=21)
Anaemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 3
Ear pain (Ear and labyrinth disorders) | 1
Euthyroid sick syndrome (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Anal incontinence (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 2
Chills (General disorders) | 4
Facial pain (General disorders) | 1
Fatigue (General disorders) | 3
General physical health deterioration (General disorders) | 1
Inflammation (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 1
Pyrexia (General disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1
Graft versus host disease in skin (Immune system disorders) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Colonic abscess (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Moraxella infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Blood creatinine decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Blood sodium decreased (Investigations) | 1
Drug level fluctuating (Investigations) | 1
Immunosuppressant drug level decreased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Spleen scan abnormal (Investigations) | 1
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Scrotal dermatitis (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Subclavian vein thrombosis (Vascular disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT04240886/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04240886/SAP_001.pdf